CLINICAL TRIAL: NCT04536506
Title: Comparison of the Effectiveness of Bobath Therapy and Vojta Technique in Babies With Down Syndrome Aged 0-24 Months: A Randomized Controlled Study
Brief Title: Bobath and Vojta Therapy for DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYŞE ÜNAL, Research assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/66911
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Down Syndrome; Motor Performance; Bobath Therapy; Vojta Technique
Keywords: infant with Down Syndrome; Bobath therapy; Vojta technique
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Bobath group received 45 min of sessions three times weekly for 12 weeks.
  Interventions: Other: Bobath Therapy
- Control group (Active Comparator): Vojta group received the following three times weekly for 12 weeks.
  Interventions: Other: Vojta technique

INTERVENTIONS:
Other: Bobath Therapy — Bobath group received 45 min of sessions three times weekly for 12 weeks. An individual program was scheduled for each case following pre-assessment. It was targeted to enable normal posture, facilitation of corrective balance and protective responses and development of normal movement patterns
  Arms: Treatment group
Other: Vojta technique — Vojta group received the following three times weekly for 12 weeks: 1. Reflex crawling, 2. First stage of reflex turning, 3. Second stage of reflex turning. Stimuli (pressure and stretch) for 30-60 sec were given by using the main stimulus points and auxiliary stimulus points together.
  Arms: Control group

SUMMARY:
Different physiotherapy approaches and education programs are applied to minimize motor and mental impairment in children with Down syndrome (DS). The present study was conducted with the aim of comparing the effectiveness of two different physiotherapy approaches in babies with Down syndrome in the early period.

A total of 23 babies with DS aged between 0-24 months were included in the study. Infants were randomly divided to two groups: Bobath therapy (BT) group included 12 infants (6 girls and 6 boys) and Vojta technique (VT) group included 11 infants (4 girls and 7 boys). The infants were applied a total of 12 sessions of physiotherapy (twice weekly during 6 weeks). Alberta Infant Motor Scale (AIMS) was used for comparison of motor development level before and after the therapy. Emotional status of the mothers was evaluated with Beck Depression Scale (BDS) and quality of life was evaluated with Nottigham Health Profile (NHP).

ELIGIBILITY:
Inclusion Criteria:

* being between 0 and 2 years
* being diagnosed with DS

Exclusion Criteria:

* having an additional neuro-motor disease

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
Alberta Infant Motor Scale | 12 weeks
  Alberta Infant Motor Scale is a tool which evaluates the infants from baby to independently walking children and measures delay in motor performance, enables families and clinicians to obtain data about motor performance of the infant, compares motor performance before and after therapy. The child is observed when performing spontaneous behaviors with a certain postural control. The scale measures weight transfer, posture and anti-gravity movements at supine, prone, sitting and standing positions with 58 items. The child receives 1 point for the movements he/she can perform and 0 point for the ones that he/she cannot perform. It is a reliable test with norm reference and suitable for clinical use due to taking short time.

SECONDARY OUTCOMES:
Beck Depression Scale | 12 weeks
  Beck Depression Scale is a scale used for evaluating emotional status of the mothers and it was arranged so as to include the symptoms of depression. Items of the scale were prepared based on clinical observations and data, not based on any hypothetical opinion. The Likert type scale is composed of 21 symptom categories. Each symptom category is scored between 0 and 3 with the highest possible score of 63. Higher scores indicates more severe depression.
Nottingham Health Profile | 12 weeks
  Nottingham Health Profile was used for assessment of quality of life of the mothers. This is a scale which is commonly used in clinical practice and includes 38 items that evaluate quality of life in 6 sections (pain, energy level, social isolation, emotional reaction, physical activity). Ratio of the "yes" answers is evaluated and each section is scored between 0 and 100 where 0 is the best and 100 is the worst score

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No